CLINICAL TRIAL: NCT04809935
Title: Endoscopic Ultrasound Guided Coeliac Plexus Block Versus Radiofrequency Ablation in Pain Relief of Patients With Intractable Pain Due to Malignancy A Randomized Controlled Study
Brief Title: EUS-Coeliac Plexus Block Versus Radiofrequency Ablation in Pain Relief of Patients With Malignancy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Ma Ka Wing, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 204610401
Record Dates: First submitted 2021-03-10; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Cancer of Pancreas; Pancreatic Neoplasms; Pain; Cancer-Associated Pain; Pain Management
Keywords: Endoscopic Ultrasound Guided; Radiofrequency Ablation; Coeliac plexus neurolysis; Pancreatic cancer; Pain Relief; Chemical coeliac plexus neurolysis; Coeliac plexus ablation; Cancer pain
MeSH Terms: conditions — Pancreatic Neoplasms; Pain; Cancer Pain; Agnosia | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- EUS-CPB (Active Comparator): Chemical ablation of the coeliac plexus
  Interventions: Drug: 98% dehydrated alcohol
- EUS-CPA (Active Comparator): Radiofrequency ablation of the coeliac plexus
  Interventions: Device: 19G EUSRA needle, Taewoong Medical, Korea

INTERVENTIONS:
Drug: 98% dehydrated alcohol — * coeliac plexus is identified and punctured
  * Injection of 10 mL of .25% bupivacaine, followed by 10 mL of 98% dehydrated alcohol.
  Other Names: Chemical Ablation
  Arms: EUS-CPB
Device: 19G EUSRA needle, Taewoong Medical, Korea — * 10W-30W RFA will be applied unilaterally or bilaterally depends on individual anatomical characteristics for 10-50s
  * Complete ablation of coeliac plexus nervous tissue is confirmed by appearance of air-bubble ultrasound scan
  Arms: EUS-CPA

SUMMARY:
Many cancer patients suffer from intractable pain and which is often suboptimally controlled by even strong opioid analgesics. Coeliac plexus neurolysis (CPN) is procedure which intended to permanently destroy the nociceptive pathway that transmits the pain caused by the tumour. It can be with different approaches, such as percutaneously guided by fluoroscopy, echo-endoscopically or surgically with endoscopic approach being the more popular one in many centers equipped with echo-endoscopic services. The effect of CPN has been well established by some retrospective series. The overall response rate to CPN ranges from 70-90%, however, the analgesic effect is limited and up to roughly around 3 months. It is believed that the short-lasting analgesic effect is related to incomplete neurolysis by absolute alcohol injection.

Recently, radiofrequency ablation (RFA) of coeliac plexus has been introduced as another mode of CPN. So far, only one small single center randomized controlled trial (RCT) suggesting superior performance in favour to CPN using RFA. This result has to be validated and by a RCT with larger sample size. In addition, data concerning the quality of life (QOL) improvement and cost-effectiveness need to be further elucidated. Therefore, the aim of this study is to perform a RCT to look into these issues.

DETAILED DESCRIPTION:
The aim of this study is to compare the efficacy of EUS-guided CPN versus radiofrequency ablation in patients with pain related to pancreatic cancer. By performing a randomized controlled trial, the clinical outcomes and cost-effectiveness of this new RFA treatment approach can be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 year-old
* Patients who give informed consent to the study
* Suboptimal pain control with regular analgesics
* Inoperable cancer of pancreas

Exclusion Criteria:

* Patients who refuse to give consent
* Patients aged <18 years
* EUS not possible due to:

Problem related to scope insertion such as trismus, stenosis of the upper GI tract Coagulopathy with INR >1.5 or platelet count < 70

* Low oxygen saturation or extreme blood pressure render endoscopic procedure unsafe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Pain score | 4 weeks
  Pain score at 4 weeks after procedure (by VAS score)

SECONDARY OUTCOMES:
Technical success rate | 2 weeks, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  Technical success rate
Clinical success rate | 2 weeks, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  Decrease of pain level by 30% from pre-procedural baseline
Duration of procedure | Up to 1 hour
  Time from injection of pre-medication to procedure last observation recording at the procedure suite
Time to pain score drop by 50% | Through study completion, an average of 2 year
  Time to Visual Analog Score drop by 50%
Short term complication rate | Up to 1 week
  Complication rate
Long term complication rate | Through study completion, an average of 2 year
  Complication rate
Hospital length of stay | Up to 100 months
  Hospital length of stay
Health status (Quality of life) | 2 weeks, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  The Short Form (36) Health Survey
Quality of life (QOL) in patients with pancreatic cancer | 2 weeks, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  PAN-26 questionnaire
Quality of life (QOL) of cancer patients | 2 weeks, 4 weeks, 8 weeks, 12 weeks, 24 weeks
  QLQ-C30 questionnaire
Cost-effectiveness of two types approach | Through study completion, an average of 2 year
  Total cost ($) of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ka Wing Ma, MBBS, MS, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong